CLINICAL TRIAL: NCT05999747
Title: A Phase 3, Multicenter, Prospective, Randomized, Open-label Study for Intraoperative Ureter(s) Visualization When Using ASP5354 With Near-infrared Fluorescence (NIR-F) Imaging in Adult Participants Undergoing Minimally Invasive and Open Abdominopelvic Surgeries
Brief Title: A Study to Find Out if ASP5354 Can Clearly Help Show the Ureter During Surgery in People With or Without Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5354-CL-0303
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Intraoperative Ureter Visualization; Abdominolpelvic Surgery
Keywords: ASP5354; Pudexacianinium chloride; Latrogenic ureteral injury; Abdominopelvic surgery; Near-infrared Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- White Light/near-infrared fluorescence - Adults with normal renal function or mild renal impairment (Experimental): Adult participants with normal renal function or mild renal impairment will receive a single dose of ASP5354
  Interventions: Drug: pudexacianinium chloride
- White Light - Adults with normal renal function or mild renal impairment (Experimental): Adult participants with normal renal function or mild renal impairment will receive a single dose of ASP5354
  Interventions: Drug: pudexacianinium chloride
- White Light/near-infrared fluorescence - Adults with moderate or severe renal impairment (Experimental): Adult participants with moderate or severe renal impairment will receive a single dose of ASP5354
  Interventions: Drug: pudexacianinium chloride

INTERVENTIONS:
Drug: pudexacianinium chloride — Intravenous
  Other Names: ASP5354

SUMMARY:
The ureter is the tube that carries urine from the kidneys to the bladder. It is difficult for surgeons to see the ureter during abdominal surgery. This could lead to injuring the ureter which, although rare, could be serious.

This study is about a potential new medical dye, called ASP5354. This dye is injected into the person at the start of surgery and is detected in the ureter. This is done by an imaging machine which has an option called near infrared fluorescence, or NIR-F. Together they show live images of specific parts of the body. In this study, ASP5354 is used with an imaging machine with a NIR-F option to show live images of the ureter during surgery.

People with kidneys that work properly and those with kidney problems can take part in this study. The main goal of the study is to find out how clearly the ureter can be seen with ASP5354 during surgery in people whose kidneys work properly or who have mild kidney problems. To do this, the surgeons will inject ASP5354 into the person having surgery. Then, the surgeons will compare images of the ureter with an imaging machine using normal white light and with the NIR-F option. Imaging using normal white light is the standard way surgeons see the ureter during surgery.

People 18 years or older, with or without kidney disease, who were going to have certain abdominal surgeries may be able to take part.

Everyone taking part will receive ASP5354 during surgery, but how the imaging is done will depend on which group they are in. Before surgery, the people whose kidneys work properly or who have mild kidney problems will be assigned into 1 of 2 groups by chance alone. Images of the ureter will be checked in 1 group using normal white light and the other group using normal white light and NIR-F. People with more severe kidney problems will not be assigned to 1 of 2 groups: all images of the ureter will be checked using normal white light and NIR-F.

At the start of surgery, the surgeon will inject ASP5354 into the person having surgery, then will start recording a video of the surgery. Then, after 30 minutes, the surgeon will record how well the ureter can be seen. This will be done by either using normal white light, or normal white light and NIR-F, depending on which group each person having surgery is assigned. For the group to be checked with normal white light and NIR-F, the surgeon will do this check every 30 minutes until the end of surgery. For the group to be checked with normal white light only, the surgeon will only do this check after the first 30 minutes. A group of medical experts will also record how well the ureter can be seen in the surgery videos. The medical experts will not be directly involved in this study. They won't know who the images belong to or which group they are from.

During the study, people will visit the study hospital 3 times. The first visit is to check if they can take part in the study. People will be asked about their medical history, have a medical examination, and their vital signs checked (blood pressure and pulse rate). Also, they will have some blood and urine tests. For women this may include a pregnancy test. People will have their surgery at the second visit. This will be within 28 days or 56 days of their first visit, depending on how severe their kidney problems are. This includes having some blood and urine tests before, during, and after surgery. Also, they will have a medical examination, an electrocardiogram (ECG) to check their heart rhythm, and have their vital signs checked. After surgery, people will return to the clinic 10 days later for a final check-up. They will be asked if they have had any medical problems. Also, they will have a medical examination, have their vital signs checked, and have blood and urine tests.

ELIGIBILITY:
Inclusion Criteria:

* Participant is scheduled to undergo minimally invasive or open abdominopelvic surgery that may require ureter identification
* Participant has normal renal function or has varying degrees of chronic kidney disease as defined by the National Kidney Foundation and calculated by individual estimated glomerular filtration rate (eGFR) using the modification of diet in renal disease formula

  * Adult normal/mild eGFR cohort: eGFR ≥ 60 mL/min
  * Adult moderate/severe eGFR cohort: eGFR ≥ 15 to < 60 mL/min
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential
  * Woman of childbearing potential who agrees to follow the contraceptive guidance from the time of informed consent through at least 30 days after study intervention administration.
* Female participant must agree not to breastfeed starting at the administration of ASP5354 through 30 days after ASP5354 administration.
* Female participant must not donate ova starting at the administration of ASP5354 through 30 days after ASP5354 administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception through at least 30 days after ASP5354 administration.
* Male participant must not donate sperm starting at the administration of ASP5354 through 30 days after ASP5354 administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy from the start of ASP5354 administration through 30 days after ASP5354 administration.
* Participant agrees not to participate in another interventional study involving unapproved study medications while participating in the present study.

Exclusion Criteria:

* Participant has any physical or psychiatric condition, which makes the participant unsuitable for study participation.
* Participant is anticipated to require ureteral stenting during surgery.
* Participant has an active urinary tract infection requiring antibiotic therapy.
* Participant has moderate to severe cardiac disease that limits daily functioning (New York Heart Association Class III to IV) or other medical conditions would impact safety or study compliance.
* Participant has any clinically relevant laboratory abnormality that could contraindicate surgery.
* Participant has a known or suspected hypersensitivity to ASP5354, indocyanine green (ICG) or any components of the formulation used.
* Participant has had previous exposure to ASP5354.
* Participant has been administered ICG or other NIR-F imaging agents within 48 hours prior to ASP5354 administration, with the exception of participants who receive ICG for lymphatic mapping before the surgery.
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to randomization.
* Participant is on hemodialysis, hemodiafiltration or peritoneal dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Intra-participant comparison in ureter conspicuity for white light (WL) versus near -infrared fluorescence (NIR F) at the first time point for participants with normal renal function or mild renal impairment. | Up to 45 minutes after ASP5354 administration (Day 1)
  Conspicuity will be scored individually for each illumination mode using the 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)

SECONDARY OUTCOMES:
Intra-participant comparison of ureter conspicuity scores for the WL at the first time point versus the average of all NIR-F time points for participants with normal renal function or mild renal impairment | Up to end of surgery (Day1)
  Conspicuity will be scored individually for each illumination mode using the 5-Point Likert Scale, ranging from1 (None) to 5 (Excellent)
Intra-participant comparison of ureter conspicuity scores for WL timepoint versus the end of surgery score with NIR-F for participants with normal renal function or mild renal impairment | Up to end of surgery (Day1)
  Conspicuity will be scored individually for each illumination mode using the 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Quantification of ureter conspicuity for WL and NIR-F illumination modes for all participants | Up to end of surgery (Day1)
  Ureter conspicuity will be quantified by image analysis measuring the color contrast when ASP5354 is present in the ureter.
Intra-participant difference in ureter conspicuity for WL versus NIR-F at the first time point for participants with moderate or severe renal impairment | Up to 45 minutes after ASP5354 administration (Day 1)
  Conspicuity will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Intra-participant comparison of ureter conspicuity scores for WL at the first time point versus the average of all NIR-F scores for participants with moderate or severe renal impairment | Up to end of surgery (Day1)
  Conspicuity will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Intra-participant comparison of ureter conspicuity scores for the WL at the first time point versus the end of surgery scores with NIR-F for participants with moderate or severe renal impairment | Up to end of surgery (Day1)
  Conspicuity will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Intra-participant difference in ureter conspicuity for WL versus NIR-F at the first time point for participants in all cohorts | Up to 45 minutes after ASP5354 administration (Day 1)
  Conspicuity will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Intra-participant comparison of ureter conspicuity scores for the WL at the first time point versus the average of all NIR-F time points for participants in all cohorts | Up to end of surgery (Day1)
  Conspicuity will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Intra-participant comparison of ureter conspicuity scores for the WL at the first time point versus the end of surgery score with NIR-F for participants in all cohorts | Up to end of surgery (Day1)
  Conspicuity will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Percentage of participants with an average index ureter conspicuity over all NIR-F time points at least 1 point higher than the average index ureter conspicuity over all WL time points | Up to the end of surgery (Day 1)
  Conspicuity will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Number of participants with an average index ureter conspicuity over all NIR-F time points at least 1 point higher than the average index ureter conspicuity over all WL time points | Up to the end of surgery (Day 1)
  Conspicuity will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Percentage of participants with an average index ureter conspicuity over all NIR-F time points at least 2, 3 or 4 points higher than the average index ureter conspicuity over all WL time points | Up to the end of surgery (Day 1)
  Conspicuity will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Number of participants with an average index ureter conspicuity over all NIR-F time points at least 2, 3 or 4 points higher than the average index ureter conspicuity over all WL time points | Up to the end of surgery (Day 1)
  Conspicuity will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Number of participants with Treatment-emergent adverse events (TEAEs) | Up to Day 25
  Adverse events (AEs) will be coded using MedDRA. An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A TEAE is defined as an AE observed after administration of the study intervention and up to the follow-up period.
Number of participants with serious TEAEs | Up to Day 25
  A Serious Adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or other medically important event. A serious TEAE is defined as an SAE observed after administration of the study intervention and up to the follow-up period.
Number of participants with laboratory value abnormalities and/or AEs | Up to Day 25
  Number of participants with potentially clinically significant laboratory values
Number of participants with vital sign abnormalities and/or AEs | Up to Day 25
  Number of participants potentially clinically significant vital signs
Number of participants with electrocardiogram (ECG) /cardiac monitoring abnormalities and/or AEs | Up to Day 2
  Number of participants potentially clinically significant ECGs/cardiac monitoring
Pharmacokinetics (PK) of ASP5354 in plasma: concentration | Up to 45 minutes after ASP5354 administration (Day 1)
  Concentration will be recorded from the PK plasma samples collected
Pharmacokinetics (PK) of ASP5354 in plasma: concentration | Up to the end of surgery (Day 1)
  Concentration will be recorded from the PK plasma samples collected
PK of ASP5354 in urine: concentration | Up to end of surgery (Day 1)
  Concentration will be recorded from the PK urine samples collected
PK of ASP5354 in urine: amount of ASP5354 excreted in urine (Ae) | Up to end of surgery (Day1)
  Ae will be recorded from the PK urine samples collected
PK of ASP5354 in urine: percentage of ASP5354 dose excreted into urine (Ae percentage) | Up to end of surgery (Day 1)
  Ae percentage will be recorded from the PK urine samples collected
Intra-participant difference in ureter conspicuity for WL versus NIR-F at the first time point for participants with normal renal function or mild renal impairment | Up to 45 minutes after ASP5354 administration (Day 1)
  BICR's (blinded independent central review) conspicuity assessment of the ureter will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Intra-participant comparison of ureter conspicuity scores for the WL at the first time point versus the average of all NIR-F time points for participants with normal renal function or mild renal impairment | Up to the end of surgery (Day 1)
  BICR's conspicuity assessment of the ureter when using ASP5354 with NIR-F for the duration of the surgical procedure will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Intra-participant comparison of ureter conspicuity scores for the WL at the first time point versus the end of surgery time point score with NIR-F for adults with normal renal function or mild renal impairment | Up to the end of surgery (Day 1)
  BICR's conspicuity assessment of the ureter when using ASP5354 with NIR-F for the duration of the surgical procedure will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Intra-participant difference in ureter conspicuity for WL versus NIR-F at the first time point for participants with moderate or severe renal impairment | Up to 45 minutes after ASP5343 administration (Day 1)
  BICR's conspicuity assessment of the ureter at the first time point will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Ureter conspicuity scores for the WL at the first time point versus the average of all NIR-F time points for participants with moderate or severe renal impairment | Up to the end of surgery (Day 1)
  BICR's conspicuity assessment of the ureter when using ASP5354 with NIR-F for the duration of the surgical procedure will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Ureter conspicuity scores for the WL at the first time point versus the end of surgery time point score with NIR F for participants with moderate or severe renal impairment | Up to the end of surgery (Day 1)
  BICR's conspicuity assessment of the ureter when using ASP5354 with NIR-F for the duration of the surgical procedure will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Intra-participant difference in ureter conspicuity for WL versus NIR-F at the first time point for all participants in all cohorts | Up to 45 minutes after ASP5354 administration (Day 1)
  BICR's conspicuity assessment of the ureter when using ASP5354 with NIR-F for the duration of the surgical procedure will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Ureter conspicuity scores for the WL at the first time point versus the average of all NIR-F time points for participants in all cohorts | Up to the end of surgery (Day 1)
  BICR's conspicuity assessment of the ureter when using ASP5354 with NIR-F for the duration of the surgical procedure will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Ureter conspicuity scores for the WL at the first time point versus the end of surgery time point score with NIR F for participants in all cohorts | Up to the end of surgery (Day 1)
  BICR's conspicuity assessment of the ureter when using ASP5354 with NIR-F for the duration of the surgical procedure will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Intra-participant difference in ureter conspicuity for WL versus NIR-F at the first time point by each BICR reader for participants with normal renal function or mild renal impairment | Up to 45 minutes after ASP5354 administration (Day 1)
  BICR's conspicuity assessment of the ureter will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
Concordance Correlation Coefficient (CCC), the inter-rater reliability between the investigators and BICR for the WL versus NIR-F at the first time point for participants with normal renal function or mild renal impairment | Up to 45 minutes after ASP5354 administration (Day 1)
  Determine degree of concordance between investigator's intra-operative conspicuity assessment of the ureter and BICR assessment
Intra-participant difference in ureter conspicuity for WL at the first time point versus the average of all NIR-F time points by each BICR reader for participants with normal renal function or mild renal impairment | Up to the end of surgery (Day 1)
  BICR's conspicuity assessment of the ureter will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
CCC, the inter-rater reliability between the investigators and BICR for the WL at the first timepoint versus the average of all NIR-F time points for participants with normal renal function or mild renal impairment | Up to the end of surgery (Day 1)
  Determine degree of concordance between investigator's intra-operative conspicuity assessment of the ureter and BICR assessment
Intra-participant difference in ureter conspicuity for WL at the first time point versus the end of surgery time point score with NIR-F by each BICR reader for participants with normal renal function or mild renal impairment | Up to the end of surgery (Day 1)
  BICR's conspicuity assessment of the ureter will be scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 (None) to 5 (Excellent)
CCC, inter-rater reliability between the investigators and BICR for the WL at the first time point versus the end of surgery time point score with NIR-F for participants with normal renal function or mild renal impairment | Up to the end of surgery (Day 1)
  Determine degree of concordance between investigator's intra-operative conspicuity assessment of the ureter and BICR assessment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development, Inc.
Locations (12):
- United States (12):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of South Florida, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Washington University Center, St Louis, Missouri
  - University of Nevada, Las Vegas, Las Vegas, Nevada
  - Duke University Hospital, Durham, North Carolina
  - Firsthealth of the Carolinas INC, Pinehurst, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Benaroya Research Institute at VA Mason, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/